CLINICAL TRIAL: NCT05739461
Title: The Effect of Triangular Cross-section Neck Design on Crestal Bone Stability in the Anterior Mandible: A Retrospective Study With a 5-year Follow-up
Brief Title: The Effect of Triangular Neck Design on Crestal Bone Loss
Status: Completed | Type: Observational
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Berkay Tokuç, Assist. Prof., Kocaeli University
Other Study IDs: 2022/158
Record Dates: First submitted 2023-02-12; First posted 2023-02-22 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Dental Implant Failed
Keywords: : buccal bone thickness; crestal bone loss; neck design; peri-implant soft tissue; triangular cross-section neck
MeSH Terms: interventions — Dental Implants

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- triangular cross-section neck implant
  Interventions: Other: Dental implant
- round cross-section neck implant
  Interventions: Other: Dental implant

INTERVENTIONS:
Other: Dental implant — Dental implants with triangular cross-section neck design

SUMMARY:
The objective of this retrospective study with 5-year follow-up was to compare crestal bone loss (CBL) and buccal bone thickness (BBT) around triangular cross-section neck (TN) to round neck (RN) implants retaining mandibular overdentures, using cone-beam computed tomography

DETAILED DESCRIPTION:
CBL is a multifactorial entity including factors related to patients, surgical technique, prosthetic interventions, and implant design. Thus, new developments in implant micro- and macro-features, such as modifications of surface characteristics and chemistry, type of abutment connection, thread design, and neck design have been introduced over time parallel to recent advances in implantology not only for reducing CBL, but also for preserving buccal bone dimensions around implant. Furthermore, implant neck properties have been considered as a determinant factor involved in maintenance of crestal bone around implant in various trials. Nevertheless, there is no consensus with respect to the design of implant neck for reducing CBL.

The most common implant neck design is the circular one; recently, however, a newly designed implant with a triangular neck (TN) portion was introduced, which has reduction in the neck portion on three sides. This neck design provides compression-free area to alveolar crest during implant insertion to minimize CBL. In addition, TN design also would enhance the BBT by increasing the space between the flat part of the triangle and the buccal bone cortex. Based our previous study with one-year follow-up, despite the implants with novel neck design showed a better crestal bone preservation compared to conventional neck design, long-term clinical trials determining the effect of TN are missing for validating the success of this new design. Unfortunately, the data derived from only very few short-term comparative clinical trials to date do not provide an answer on benefits of TN design over the CN implants regarding preserving crestal bone level.

Thus, this retrospective study with up-to-x-month follow-up aimed to compare CBL and BBT around implants with TN and RN retaining mandibular overdentures. The null hypothesis was that there was a difference in CBL and BBT between two implant designs in the long-term follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old.
* Mandibular total edentulism.
* Presence of sufficient residual bone width (>5 mm) and length (>10 mm).
* Sufficient keratinized gingiva crestally (≥4 mm).
* Sufficient interarch space.
* Sufficient vestibular depth.
* Patients had their teeth extracted at least three months before surgery.

Exclusion Criteria:

* Patients with any systemic disease or condition that can/could compromise osteointegration (cancer, diabetes mellitus, osteopo- rosis, and cardiovascular diseases).
* Presence of any drug use that could affect bone metabolism.
* Presence of immunocompromising conditions.
* Presence of any pathology in the mandible.
* Allergy to any drugs used in the postoperative period.
* Patients who are smokers.

Ages: 59 Years to 72 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healty patients who was inserted dental implants with two different designs
Sampling Method: Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2022-09-22 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
comparison of crestal bone loss | February 2023
comparison of buccal bone thickness | February 2023

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli University, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided